CLINICAL TRIAL: NCT06222827
Title: A Bicentric, Randomized, Double Blind, Placebo-controlled Pilot Study to Evaluate the Efficacy and Safety of Satralizumab in FSHD1
Brief Title: Study to Evaluate the Efficacy and Safety of Satralizumab in FSHD1
Acronym: REINFORCE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22-PP-24
Record Dates: First submitted 2023-12-15; First posted 2024-01-25 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Facioscapulohumeral Muscular Dystrophy 1

STUDY DESIGN:
Intervention Model Description: First period: two groups of patients who receive either satralizumab, or placebo. Second period: all patients receive satralizumab
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group of patients who receive satralizumab (Experimental)
  Interventions: Drug: Satralizumab Prefilled Syringe
- Group of patients who receive placebo (Placebo Comparator)
  Interventions: Drug: Placebo Comparator

INTERVENTIONS:
Drug: Satralizumab Prefilled Syringe — Satralizumab is supplied as prefilled syringe with 1 millimeter of solution for subcutaneous injection corresponding to 120mg of satralizumab. During the first period (double blind period), satralizumab will be administered at weeks 0, 2, 4 and every 4 weeks until week 48. During the second period (open label period), satralizumab will be administered at weeks 48, 50, 52 and every 4 weeks until week 96.
  Arms: Group of patients who receive satralizumab
Drug: Placebo Comparator — Placebo prefilled syringe is identical in composition to satralizumab, but does not contain the satralizumab active agent. It is identical in appearance and packaging to satralizumab. During the first period (double blind period), placebo will be administered at weeks 0, 2, 4 and every 4 weeks until week 48. During the second period (open label period), satralizumab will be administered at weeks 48, 50, 52 and every 4 weeks until week 96.
  Arms: Group of patients who receive placebo

SUMMARY:
Facioscapulohumeral muscular dystrophy (FSHD) is characterized by clinical diversity, with FSHD1 being the most common form. It is associated with a toxic gain of function of the Double homeobox 4 (DUX4) gene, leading to muscle cell death and weakness. Despite the lack of approved treatments, recent studies highlight inflammation's role in early FSHD progression, triggered by inappropriate DUX4 expression.

In understanding inflammation's pivotal role in FSHD, a study assessed serum cytokines in 100 adult FSHD1 patients. Out of the 20 cytokines examined, 10 showed significantly altered expression levels compared to healthy controls of similar age and sex. FSHD1 patients exhibited heightened levels of inflammatory cytokines and diminished anti-inflammatory cytokines, signaling chronic inflammation. Notably, Interleukin-6 (IL-6) emerged as a promising disease activity biomarker, displaying robust correlations with established clinical severity and functional scores.

Given the pathological significance of inflammation and the correlation of IL-6 levels with disease severity, the ReInForce study will explore the satralizumab, an IL6-receptor (IL6-R) antagonist, for its efficacy in specifically reducing muscle and systemic inflammation. By antagonizing IL-6R downstream signaling, satralizumab holds promise in mitigating inflammation and potentially curtailing fibrofatty degeneration in FSHD.

ELIGIBILITY:
Inclusion Criteria:

* Capable of understanding the written informed consent, and providing signed, dated, and witnessed written informed consent.
* Male or female subjects between the ages of 18 and 65 years, inclusive.
* Patient affiliated to a European social security system (Nice center only)
* Genetically confirmed diagnosis of typical FSHD1 with 1 to 9 D4Z4 repeats via assessment of the size of the D4Z4 array on chromosome 4. Genetic confirmation must be obtained before the subject screening assessments, including MRI, and before the baseline. Genetic confirmation can come from previous testing if verified with appropriate documentation from an accredited laboratory. Due to stable transmission of repeat sizes within families, subjects with a clinical diagnosis of FSHD who have a first-degree relative with a genetically confirmed diagnosis of FSHD1 may be entered into the study for screening assessments, including MRI.
* Clinical severity score of 2 to 4 (RICCI score; range 0-5), inclusive.
* Patients with a body weight of below or equal 100 kg
* On initial whole-body MRI, subjects with evidence of muscle fat replacement such that the total lean volume of muscles with an intermediate fat replacement (i.e. muscle with at least 10% of Muscle Fat Infiltration and no more than 50% of Muscle Fat Fraction) is at least 500 ml if there is only one intermediate muscle or 250 ml if there is more than one intermediate muscle.
* Subjects able to walk without support
* Willing to maintain same level of exercise (frequency and intensity) during the study.
* Willing and able to comply with scheduled visits, treatment plan, study restrictions, laboratory tests, contraceptive guidelines, and other study procedures.
* For female patients of childbearing potential: use adequate contraception during the treatment period and/or until treatment discontinuation.

Exclusion Criteria:

* History of any illness or any clinical condition that, in the opinion of the investigator, might confound the results of the study or pose an additional risk in administering study drug to the subject. This may include, but is not limited to, any major comorbidities (diabetes mellitus, cancer, severe autoimmune diseases, chronic renal failure, articular diseases that restricts exercise or participation in study assessments in the physician's opinion...), a history of relevant drug or food allergies; history of cardiovascular, respiratory, central nervous system disease; neuromuscular diseases except FSHD (e.g., myopathy, neuropathy, neuromuscular junction disorders)
* History of malignancy within the last 5 years, including solid tumors, hematologic malignancies and in situ carcinoma (except basal cell and squamous cell carcinomas of the skin, or in situ carcinoma of the cervix uteri that have been completely excised and cured)
* Subjects who are on drug(s) or supplements that may affect muscle function, as determined by the treating physician must be on a stable dose of that drug(s) or supplement for at least 3 months prior to the first dose of study drug and remain on that stable dose for the duration of the study.
* Orthopedic conditions, such as unresolved fracture or arthrosis, interfering or precluding testing of muscle function
* Contraindication to muscle MRI as per clinic standard practice
* Articular contracture limiting movements, scapular fixation or other surgeries, preceding or planned
* Any known hypersensitivity to satralizumab or any of its components and/or history of severe allergic reaction to a biologic agent (e.g., shock, anaphylactic reactions)
* Evidence of latent or active tuberculosis (TB; excluding patients receiving chemoprophylaxis for latent TB infection for at least 4 weeks prior to enrollment), active opportunistic or life-threatening infections
* History of diverticulitis or concurrent severe GI disorders (such as symptomatic diverticulosis) that, in the investigator's opinion, may lead to increased risk of complications such as GI perforation. Infection requiring hospitalization or treatment with IV anti-infective agents within 4 weeks prior to baseline visit or oral anti-infective agents within 2 weeks prior to baseline visit (Visit 1, week 0)
* Positive screen for hepatitis B surface antigen (HbsAg), antibody (anti-HbS), hepatitis C virus (HCV) antibody.
* Acute or chronic history of liver disease
* Abnormal laboratory results with: White blood cells (WBC) < 3.0x 10^9/L ; Absolute Neutrophils Counts (ANC)< 2.0x 10^9/L ; Platelet count < 10x10^4/µl ; Absolute lymphocyte count (ALC) < 0.8x 10^3/µl ; Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 1.5 times the upper limit of normal (ULN)
* Severe renal impairment (defined as a glomerular filtration rate of <30mL/min/1.73m²)
* Vaccination with live or live-attenuated vaccines within the 6 weeks prior to randomization.
* Pregnancy or lactation
* For patients of reproductive potential, a positive result from a serum pregnancy test at screening, or not willing to use reliable means of contraception (physical barrier [patient or partner] in conjunction with a spermicidal product, contraceptive pill, patch, injectable, intrauterine device or intrauterine system) during the treatment period and for at least 3 months after the last dose of study drug.
* Any current mental condition (psychiatric disorder, senility, or dementia) that, in the opinion of the investigator, may affect study compliance or prevent understanding of the aims, investigational procedures, or possible consequences of the study.
* Use of another investigational product within 6 months or 5 half-lives (whichever is longer), or currently participating in a prospective study with an investigational product, whether it concerns an experimental drug or a medical device. Note: concurrent participation in natural history studies (non-drug, non-device studies) is not allowed during the course of the study.
* Any prior treatment with any agent targeting the IL-6 inhibition pathway (e.g. tocilizumab, sarilumab), alemtuzumab treatment, total body irradiation, or bone marrow transplantation; treatment in the past 24 weeks with an anti-B-lymphocyte antigen CD20 (e.g. rituximab, ocrelizumab), eculizumab, anti-B-lymphocyte stimulator, or any other multiple sclerosis disease-modifying treatment; treatment in the past 2 years with an anti-T-cell surface glycoprotein CD4, cladribine, cyclophosphamide, or mitoxantrone; or treatment with any other investigational drug within 3 months prior to baseline. See section 4.4.4 for details on the vaccination and immunization.
* Subject, or close relative of the subject, is the investigator or a coinvestigator, research assistant, pharmacist, study coordinator, or other staff directly involved with the conduct of the study at that site.
* Patient protected by law, under guardianship or curator ship, or not able to participate in a clinical study according to the article L.1121-16 of the French Public Health Code.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2024-01-24 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
The study will evaluate the efficacy of satralizumab compared to placebo, measured by the change during the Double Blind (DB) period (week 0 to week 48) on whole body muscle MRI. | From baseline to week 48
  Based on T1-Dixon images, muscles will be evaluated on all available sections, and a composite score describing the Muscle Fat Infiltration (MFItot, in % of total muscle), Lean Muscle Volume (LMVtot in cl) and Muscle Fat Fraction (MFFtot in % of total muscles) in intermediate muscles (muscles with at least 10% of MFI and no more than 50% of MFF) Based on T2 Short T1 Inversion Recovery (STIR), muscles will be evaluated on all available sections, and a comprehensive score describing the degree of involvement was given between 0 (absence of STIR hyperintensity) and 1 (presence of area of STIR hyperintensity).
  A STIR-Magnetic Resonance Imaging (MRI) score will be calculated as the sum of the scores of involvement of the individual muscles in each patient
The study will evaluate the efficacy of satralizumab compared to placebo, measured by the change during the Double Blind (DB) period (week 0 to week 48) on RICCI clinical severity scale score. | From baseline to week 48
  The RICCI score is a 10-grade scale that accounts for the extent of weakness in various muscular regions and considers the spread of symptoms to pelvic and leg muscles. Higher scores are assigned to subjects with involvement of pelvic and proximal lower limb muscles.
The study will evaluate the efficacy of satralizumab compared to placebo, measured by the change during the Double Blind (DB) period (week 0 to week 48) on Reachable Work Space (RWS) results with and without weights. | From baseline to week 48
The study will evaluate the efficacy of satralizumab compared to placebo, measured by the change during the Double Blind (DB) period (week 0 to week 48) on muscle strength, determined by quantitative isometric dynamometry | From baseline to week 48
The study will evaluate the efficacy of satralizumab compared to placebo, measured by the change during the Double Blind (DB) period (week 0 to week 48) on FSHD-Composite Outcome Measure (FSHD-COM) total score, sub-scale scores and individual items. | From baseline to week 48
  The FSHD Composite Outcome Measure (FSHD-COM) is an evaluator-administered scale, specifically developed for FSHD. This instrument is comprised from several independent functional tests which, when combined, give an overall score by body region, including leg, shoulder and arm, trunk, hand and balance. The lower the score is the less affected the patient is.
The study will evaluate the efficacy of satralizumab compared to placebo, measured by the change during the Double Blind (DB) period (week 0 to week 48) on FSHD-Rasch-built overall disability scale (FSHD-RODS) total score | From baseline to week 48
  The FSHD-Rasch-built overall disability scale (FSHD-RODS) is a patient-reported disease-specific interval measure suitable for detecting activity and participation restrictions in patients with FSHD. The 32-item FSHD-RODS demonstrated good discriminative validity when correlated with the MFM and an excellent test-retest reliability scores for item hierarchy and patient abilities.
The study will evaluate the efficacy of satralizumab compared to placebo, measured by the proportion of participants with an improvement in the FSHD Patient Global Impression of Change scale (FSHD-PGIC) during the Double Blind period (week 0 to week 48) | From baseline to week 48
  The self-report measure FSHD-Patient Global Impression of Change (FSHD-PGIC) reflects a patient's belief about the efficacy of treatment. PGIC is a 7-point scale depicting a patient's rating of overall improvement. Patients rate their change as: Very much improved (1), Much improved (2), Minimally improved (3), No change (4), Minimally worse (5), Much worse (6), Very much worse (7).
The study will evaluate the efficacy of satralizumab compared to placebo, measured by the proportion of participants with an improvement in FSHD Clinical Global Impressions of Change scale (FSHD-CGIC) during the Double Blind period (week 0 to week 48) | From baseline to week 48
  The physician-report measure FSHD-Clinical Global Impression of Change (FSHD-CGIC) asked to the clinicians to rate the degree of change observed in a patient since the beginning of the study. CGIC is a 7-point scale and physicians rate patients change as: Very much improved (1), Much improved (2), Minimally improved (3), No change (4), Minimally worse (5), Much worse (6), Very much worse (7).
The study will evaluate the efficacy of satralizumab compared to placebo, measured by the change during the Double Blind (DB) period (week 0 to week 48) on the number of falls reported. | From baseline to week 48
The study will evaluate the efficacy of satralizumab compared to placebo, measured by the change during the Double Blind (DB) period (week 0 to week 48) on Neuromuscular Disease Independence Scale-Upper Limb Module (NMDIS-ULM) total score | From baseline to week 48
  The Neuromuscular Disease Independence Scale-Upper Limb Module (NMDIS-ULM) is an adaptation of the SMA Independence Scale-Upper Limb Module (SMAIS-ULM) which have been developed to measure the level of assistance required for activities related to upper limb function. Higher score are assigend to subject requiring help in daily activities.
The study will evaluate the efficacy of satralizumab compared to placebo, measured by the change during the Double Blind (DB) period (week 0 to week 48) on Neuromuscular Disease Independence Scale-Ambulatory (NMDIS-Amb) total score. | From baseline to week 48
  The Neuromuscular Disease Independence Scale-Ambulatory (NMDIS-Amb) is an adaptation of the SMA Independence Scale Ambulatory module (SMAIS-Amb) which have been developed to measure the level of assistance required for activities related to motor function. Higher score are assigned to subjects unable to perform the activity present in the questionnaire
The study will evaluate the efficacy of satralizumab compared to placebo, measured by the change during the Double Blind (DB) period (week 0 to week 48) on inflammation, and specifically on molecular biomarkers associated with inflammation. | From baseline to week 48
  A recent study has investigated the level of 20 inflammatory cytokines to determine severity biomarker in FSHD. Among the 20 tested cytokines, 10 of them displayed a significantly different expression level between patients and control. In the present study, the efficacy of satralizumab versus placebo to reduce the inflammatory cytokines production will be investigated by comparing the change from baseline in the molecular biomarkers associated with inflammation. Biomarkers will include, but are not limited to the following:
  * Serum IL-6, sIL-6R measured by Quantikine ELISA, from R&D System, CRP,
  * Molecular biomarkers associated with inflammation such as IFN-γ, IL-1β, TNF-α, VEGF, IL1-RA, IL-6-R, sICAM-1, sVCAM-1 and SAA, measured by V-PLEX assays (MesoScale Discovery).
The study will evaluate the safety and tolerability of satralizumab compared to placebo, measured by the type, frequency, severity, seriousness, and relationship of Adverse Events to satralizumab during the Double Blind (DB) period (week 0 to week 48). | From baseline to week 48
The study will evaluate the safety and tolerability of satralizumab compared to placebo, measured by the incidence of Adverse events of special interest (AESIs) and selected AEs during the Double Blind (DB) period (week 0 to week 48). | From baseline to week 48
The study will evaluate the safety and tolerability of satralizumab compared to placebo, measured by the number of subjects discontinuing study drug due to an AE during the Double Blind (DB) period (week 0 to week 48). | From baseline to week 48
The study will evaluate safety and tolerability of satralizumab compared to placebo, measured by frequency of clinically significant changes from baseline in laboratory test, vital signs, and physical examination results during the Double Blind period | From baseline to week 48

SECONDARY OUTCOMES:
The study will evaluate the efficacy of satralizumab compared to placebo, measured by the change during Double Blind (DB) and Open-label (OL) periods (week 0 to week 96) on whole body muscle MRI. | From baseline to week 96
  Based on T1-Dixon images, muscles will be evaluated on all available sections, and a composite score describing the Muscle Fat Infiltration (MFItot, in % of total muscle), Lean Muscle Volume (LMVtot in cl) and Muscle Fat Fraction (MFFtot in % of total muscles) in intermediate muscles (muscles with at least 10% of MFI and no more than 50% of MFF) Based on T2 Short T1 Inversion Recovery (STIR), muscles will be evaluated on all available sections, and a comprehensive score describing the degree of involvement was given between 0 (absence of STIR hyperintensity) and 1 (presence of area of STIR hyperintensity).
  A STIR-Magnetic Resonance Imaging (MRI) score will be calculated as the sum of the scores of involvement of the individual muscles in each patient
The study will evaluate the efficacy of satralizumab compared to placebo, measured by the change during Double Blind (DB) and Open-label (OL) periods (week 0 to week 96) on RICCI clinical severity scale score | From baseline to week 96
  The RICCI score is a 10-grade scale that accounts for the extent of weakness in various muscular regions and considers the spread of symptoms to pelvic and leg muscles. Higher scores are assigned to subjects with involvement of pelvic and proximal lower limb muscles.
The study will evaluate the efficacy of satralizumab compared to placebo, measured by the change during Double Blind (DB) and Open-label (OL) periods (week 0 to week 96) on Reachable Work Space (RWS) results with and without weights. | From baseline to week 96
The study will evaluate the efficacy of satralizumab compared to placebo, measured by the change during Double Blind (DB) and Open-label (OL) periods (week 0 to week 96) on muscle strength, determined by quantitative isometric dynamometry | From baseline to week 96
The study will evaluate the efficacy of satralizumab compared to placebo, measured by the change during Double Blind and Open-label periods on FSHD-Composite Outcome Measure (FSHD-COM) total score, sub-scale scores and individual items | From baseline to week 96
  The FSHD Composite Outcome Measure (FSHD-COM) is an evaluator-administered scale, specifically developed for FSHD. This instrument is comprised from several independent functional tests which, when combined, give an overall score by body region, including leg, shoulder and arm, trunk, hand and balance. The lower the score is the less affected the patient is.
The study will evaluate the efficacy of satralizumab compared to placebo, measured by the change during Double Blind (DB) and Open-label (OL) periods (week 0 to week 96) on FSHD-Rasch-built overall disability scale (FSHD-RODS) total score | From baseline to week 96
  The FSHD-Rasch-built overall disability scale (FSHD-RODS) is a patient-reported disease-specific interval measure suitable for detecting activity and participation restrictions in patients with FSHD. The 32-item FSHD-RODS demonstrated good discriminative validity when correlated with the MFM and an excellent test-retest reliability scores for item hierarchy and patient abilities.
The study will evaluate the efficacy of satralizumab compared to placebo, measured by the proportion of participants with an improvement in the FSHD Patient Global Impression of Change scale (FSHD-PGIC) during Double Blind and Open-label periods | From baseline to week 96
  The self-report measure FSHD-Patient Global Impression of Change (FSHD-PGIC) reflects a patient's belief about the efficacy of treatment. PGIC is a 7-point scale depicting a patient's rating of overall improvement. Patients rate their change as: Very much improved (1), Much improved (2), Minimally improved (3), No change (4), Minimally worse (5), Much worse (6), Very much worse (7).
The study will evaluate the efficacy of satralizumab compared to placebo, measured by the proportion of participants with an improvement in the FSHD Clinical Global Impressions of Change scale (FSHD-CGIC) during Double Blind and Open-label periods | From baseline to week 96
  The physician-report measure FSHD-Clinical Global Impression of Change (FSHD-CGIC) asked to the clinicians to rate the degree of change observed in a patient since the beginning of the study. CGIC is a 7-point scale and physicians rate patients change as: Very much improved (1), Much improved (2), Minimally improved (3), No change (4), Minimally worse (5), Much worse (6), Very much worse (7).
The study will evaluate the efficacy of satralizumab compared to placebo, measured by the change during Double Blind (DB) and Open-label (OL) periods (week 0 to week 96) on the number of falls reported | From baseline to week 96
The study will evaluate the efficacy of satralizumab compared to placebo, measured by the change during Double Blind (DB) and Open-label (OL) periods on Neuromuscular Disease Independence Scale-Upper Limb Module (NMDIS-ULM) total score. | From baseline to week 96
  The Neuromuscular Disease Independence Scale-Upper Limb Module (NMDIS-ULM) is an adaptation of the SMA Independence Scale-Upper Limb Module (SMAIS-ULM) which have been developed to measure the level of assistance required for activities related to upper limb function. Higher score are assigend to subject requiring help in daily activities.
The study will evaluate the efficacy of satralizumab compared to placebo, measured by the change during Double Blind (DB) and Open-label (OL) periods (week 0 to week 96) on Neuromuscular Disease Independence Scale-Ambulatory (NMDIS-Amb) total score | From baseline to week 96
  The Neuromuscular Disease Independence Scale-Ambulatory (NMDIS-Amb) is an adaptation of the SMA Independence Scale Ambulatory module (SMAIS-Amb) which have been developed to measure the level of assistance required for activities related to motor function. Higher score are assigned to subjects unable to perform the activity present in the questionnaire
The study will evaluate the efficacy of satralizumab compared to placebo, measured by the change during Double Blind (DB) and Open-label (OL) periods on inflammation, and specifically on molecular biomarkers associated with inflammation | From baseline to week 96
  A recent study has investigated the level of 20 inflammatory cytokines to determine severity biomarker in FSHD. Among the 20 tested cytokines, 10 of them displayed a significantly different expression level between patients and control. In the present study, the efficacy of satralizumab versus placebo to reduce the inflammatory cytokines production will be investigated by comparing the change from baseline in the molecular biomarkers associated with inflammation. Biomarkers will include, but are not limited to the following:
  * Serum IL-6, sIL-6R measured by Quantikine ELISA, from R&D System, CRP,
  * Molecular biomarkers associated with inflammation such as IFN-γ, IL-1β, TNF-α, VEGF, IL1-RA, IL-6-R, sICAM-1, sVCAM-1 and SAA, measured by V-PLEX assays (MesoScale Discovery).
The study will evaluate the safety and tolerability of satralizumab compared to placebo, measured by the type, frequency, severity, seriousness, and relationship of Adverse Events to satralizumab during Double Blind and Open-label periods | From baseline to week 96
The study will evaluate the safety and tolerability of satralizumab compared to placebo, measured by the incidence of Adverse events of special interest (AESIs) and selected AEs during Double Blind (DB) and Open-label (OL) periods (week 0 to week 96) | From baseline to week 96
The study will evaluate the safety and tolerability of satralizumab compared to placebo, measured by the number of subjects discontinuing study drug due to an AE during Double Blind (DB) and Open-label (OL) periods (week 0 to week 96) | From baseline to week 96
The study will evaluate safety/tolerability of satralizumab versus placebo, measured by frequency of clinically significant changes from baseline in laboratory test, vital signs, and physical examination results during Double Blind and Open-label periods | From baseline to week 96

CONTACTS AND LOCATIONS:
Locations (2):
- CHEO Research Institute Ottawa, Ottawa, Ontario, Canada
- CHU de Nice, Nice, Alpes Maritimes, France

IPD SHARING:
Plan to Share IPD: No